CLINICAL TRIAL: NCT04409717
Title: Evaluation of the Long Term Efficacy of Endovascular Treatment of Type 2 Endoleaks
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Principal Investigator, Eric STEINMETZ, Professor, Centre Hospitalier Universitaire Dijon
Other Study IDs: CCVT - type 2 endoleaks
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated for type II endoleaks: Patients treated for type II endoleaks between the 01 January 2008 and the 31 March 2018 in the Cardiovascular and Thoracic Surgery Unit of Dijon Burgundy University Hospital
  Interventions: Procedure: Type II endoleak treatment

INTERVENTIONS:
Procedure: Type II endoleak treatment — Type II endoleak endovascular treatment

SUMMARY:
Endovascular treatment has become the first choice to repair abdominal aortic aneurym, but exposes patients to a risk of endoleaks. Although treatment of type 1 and 3 endoleaks has proven to prevent aneurysms from rupture, controversies remain about type 2 endoleaks. The investigators described the different techniques of type 2 endovascular repair, and their efficacy at short and long term..

ELIGIBILITY:
Inclusion Criteria:

* All patients treated for type II endoleaks by endovascular therapy

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for type II endoleaks by endovascular therapy between the 01 January 2008 and the 31 December 2018
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of type II endoleaks treated with endovascular intervention | 12 years

SECONDARY OUTCOMES:
Type of type II endoleaks treatment | 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric STEINMETZ, MD, Principal Investigator — Cardiovascular and Thoracic Surgery Unit - Dijon Univeristy Hospital
Locations (1):
- Cardiovascular and thoracic surgery unit, CHU Dijon, Dijon, France

IPD SHARING:
Plan to Share IPD: No
All patients signed a institutional form prior to the procedure stating that they did not object to the use of their medical data for research purposes.
  Before inclusion, all patients (or a trusted person) were informed about the study and its objectives. No opposition was expressed.